CLINICAL TRIAL: NCT00206648
Title: A Randomized, Rater-blinded, Multicenter, Parallel-group Study Comparing the Efficacy and Safety of Betaseron 250 µg Subcutaneously Every Other Day With Avonex 30 µg Intramuscularly Once Per Week in Relapsing-remitting Multiple Sclerosis Patients Previously Treated With Avonex
Brief Title: An Efficacy and Safety Comparison Study of Two Marketed Drugs in Patients With Relapsing-remitting MS
Acronym: ABOVE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 91293; 307245
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Interferon beta-1b

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Betaferon/Betaseron
- Arm 2 (Active Comparator)
  Interventions: Drug: Betaferon/Betaseron

INTERVENTIONS:
Drug: Betaferon/Betaseron — Betaseron 250 µg SC every other day
  Arms: Arm 1
Drug: Betaferon/Betaseron — Avonex 30 µg IM once per week
  Arms: Arm 2

SUMMARY:
The purpose of this study is to determine the difference in preventing a relapse between Betaseron and Avonex. Patients with RRMS currently treated with Avonex will be randomized into 2 equal-size arms; one arm will continue on the standard dose of Avonex; one arm will be converted to Betaseron standard dose.

DETAILED DESCRIPTION:
This study has previously been posted by Berlex, Inc. Berlex, Inc. has been renamed to Bayer HealthCare Pharmaceuticals, Inc.Bayer HealthCare Pharmaceuticals, Inc.is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* RRMS patients that are receiving treatment with Avonex 30 µg once weekly

Exclusion Criteria:

* Primary Progressive or Secondary Progressive MS

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 271 (Actual)
Dates: Start 2003-03; Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Time to onset of first relapse | Time to onset of first relapse

SECONDARY OUTCOMES:
Number of patients relapse free at week 104 | At week 104

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (51):
- United States (49):
  - Tucson, Arizona
  - Berkeley, California
  - Irvine, California
  - Loma Linda, California
  - Los Angeles, California
  - Sacramento, California
  - San Jose, California
  - Walnut Creek, California
  - Wilmington, Delaware
  - Melbourne, Florida
  - Miami, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Columbus, Georgia
  - Savannah, Georgia
  - Flossmoor, Illinois
  - Springfield, Illinois
  - Fort Wayne, Indiana
  - Indianapolis, Indiana
  - Des Moines, Iowa
  - Kansas City, Kansas
  - Shreveport, Louisiana
  - Baltimore, Maryland
  - Detroit, Michigan
  - Golden Valley, Minnesota
  - Minneapolis, Minnesota
  - Rochester, Minnesota
  - Kansas City, Missouri
  - St Louis, Missouri
  - Reno, Nevada
  - Albuquerque, New Mexico
  - Albany, New York
  - Buffalo, New York
  - Mineola, New York
  - New York, New York
  - Asheville, North Carolina
  - Winston-Salem, North Carolina
  - Dayton, Ohio
  - Oklahoma City, Oklahoma
  - Medford, Oregon
  - Philadelphia, Pennsylvania
  - Providence, Rhode Island
  - Charleston, South Carolina
  - Houston, Texas
  - Fairfax, Virginia
  - Roanoke, Virginia
  - Seattle, Washington
  - Tacoma, Washington
- Canada (2):
  - Nepean, Ontario
  - Ottawa, Ontario